CLINICAL TRIAL: NCT03265704
Title: Maternal Pregnancy Induced Hypertension and Hematological Profile of Newborns
Brief Title: Maternal High Blood Pressure and Newborn's Blood Profile
Acronym: MPIHHPN
Status: Completed | Type: Observational
Sponsor: Romanian Society of Anesthesia and Intensive Care (Other)
Collaborators: University of Medicine and Pharmacy "Victor Babes" Timisoara (Other); Timişoara County Emergency Clinical Hospital (Other)
Responsible Party: Principal Investigator, Alexandru Florin Rogobete, MSc, PhDs, Clinical Researcher, Romanian Society of Anesthesia and Intensive Care
Other Study IDs: 201601MP
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Maternal-Fetal Exchange
Keywords: Maternal PIH; Neonatal thrombocytopenia; Neonatal neutropenia
MeSH Terms: conditions — Thrombocytopenia, Neonatal Alloimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- AGA Neonates: AGA Control Group Appropriate for gestational age newborns of healthy mothers
  Interventions: Other: AGA - Control group
- SGA Neonates: SGA - Control Group Small for gestational age newborns of healthy mothers
  Interventions: Other: SGA - Control group
- AGA-PIH Neonates: AGA-PIH Study Group Appropriate for gestational age newborns of mothers with pregnancy induced hypertension
  Interventions: Other: AGA-PIH Study group
- SGA-PIH Neonates: SGA-PIH Study Group Small for gestational age newborns of mothers with pregnancy induced hypertension
  Interventions: Other: SGA-PIH Study group

INTERVENTIONS:
Other: AGA - Control group — Data processing from Patient Medical Files
  Groups: AGA Neonates
Other: SGA - Control group — Data processing from Patient Medical Files
  Groups: SGA Neonates
Other: AGA-PIH Study group — Monitoring PIH-related changes in the newborn
  Groups: AGA-PIH Neonates
Other: SGA-PIH Study group — Monitoring PIH-related changes in the newborn
  Groups: SGA-PIH Neonates

SUMMARY:
Maternal high blood pressure remodels the intrauterine environment of the fetus by altering hormonal and cellular signaling patterns and, as a result increases the risk of fetal and neonatal mortality and morbidity. Newborns of these mothers have an increased risk of intrauterine growth restriction, premature birth and hematological abnormalities, such as thrombocytopenia, polycythemia, and neutropenia. The purpose of the article is to review neonatal thrombocytopenia and neutropenia as a consequence of maternal high blood pressure and to establish the optimal management of these cases.

DETAILED DESCRIPTION:
Pregnancy induced hypertension (PIH) and preeclampsia (preE) are caused by gestation and have an onset after 20 weeks of pregnancy. Although the exact etiology of PIH and preE remains unknown, two interconnected mechanisms have been identified to play an important role in the pathogenesis: dysfunction of the placental trophoblast and endothelial dysfunction within the maternal systemic vasculature. The endothelium has been identified as the target tissue of the disease. Endothelial alterations ultimately manifest as placental hypoxia and hypoplasia. The neonatal thrombocytopenia and neutropenia after pregnancy-induced hypertension is a result of inhibition of fetal bone marrow production of the myeloid lineage due to intrauterine hypoxic environment. This study aims to investigate the hematological profile in term and preterm infants born to mothers with preeclampsia. The current retrospective observational study was conducted at the Clinic of Obstetrics, Gynecology and Neonatology of the Emergency County Hospital, Timisoara over a period of three years, from January 2014 to December 2016. All inborn patient files were analyzed as anonymised limited data sets from archived records of the Neonatology Department.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-28 days
* Newborns of healthy mothers;
* Newborns of mothers with Pregnancy Induced Hypertension;
* Inborn Patients;
* Written Informed Consent signed by legal guardian.

Exclusion Criteria:

* Maternal disease other than PIH;
* Syndromal, chromosomal or infectious diseases of the newborns;
* Causes other then PIH for perinatal asphyxia.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns admitted to the Neonatology Department who met the Inclusion Criteria.
Sampling Method: Probability Sample
Enrollment: 6108 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Hematological Changes in the Newborns of Mothers with Pregnancy Induced Hypertension | Blood profiles of newborns aged between 1-28 days were evaluated.
  Evaluating the impact of Maternal Pregnancy Induced Hypertension on fetal and neonatal hematopoiesis with focus on the myeloid lineage.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Florin Rogobete, PhDs, Principal Investigator — Romanian Society of Anesthesia and Intensive Care; Dorel Sandesc, Prof, Study Chair — Romanian Society of Anesthesia and Intensive Care; Ovidiu Bedreag, Assoc Prof, Study Director — Romanian Society of Anesthesia and Intensive Care
Locations (1):
- Romanian Society of Anesthesia and Intensive Care, Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhat YR, Cherian CS. Neonatal thrombocytopenia associated with maternal pregnancy induced hypertension. Indian J Pediatr. 2008 Jun;75(6):571-3. doi: 10.1007/s12098-008-0110-x. Epub 2008 Aug 31. PMID 18759083
- [Background] Backes CH, Markham K, Moorehead P, Cordero L, Nankervis CA, Giannone PJ. Maternal preeclampsia and neonatal outcomes. J Pregnancy. 2011;2011:214365. doi: 10.1155/2011/214365. Epub 2011 Apr 4. PMID 21547086
- [Background] de Zegher F, Francois I, van Helvoirt M, Van den Berghe G. Clinical review 89: Small as fetus and short as child: from endogenous to exogenous growth hormone. J Clin Endocrinol Metab. 1997 Jul;82(7):2021-6. doi: 10.1210/jcem.82.7.4007. No abstract available. PMID 9215266
- [Background] Christensen RD, Yoder BA, Baer VL, Snow GL, Butler A. Early-Onset Neutropenia in Small-for-Gestational-Age Infants. Pediatrics. 2015 Nov;136(5):e1259-67. doi: 10.1542/peds.2015-1638. Epub 2015 Oct 12. PMID 26459642